CLINICAL TRIAL: NCT00877591
Title: Interaction of Buprenorphine With HIV Medications and Tuberculosis Medications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: State University of New York at Buffalo (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA013004 (NIH)
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Opioid Dependency; HIV Infections
Keywords: Interaction of Buprenorphine with HIV and TB Medications
MeSH Terms: conditions — HIV Infections | interventions — fosamprenavir; Ritonavir; Darunavir; Rifampin; Rifabutin; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Buprenorphine + Fosamprenavir/Ritonavir
  Interventions: Drug: Fosamprenavir/Ritonavir; Drug: Buprenorphine
- 2 (Active Comparator): Control Fosamprenavir/Ritonavir
  Interventions: Drug: Fosamprenavir/Ritonavir
- 3 (Experimental): Buprenorphine + Darunavir/Ritonavir
  Interventions: Drug: Darunavir/Ritonavir; Drug: Buprenorphine
- 4 (Active Comparator): Control Darunavir/Ritonavir
  Interventions: Drug: Darunavir/Ritonavir
- 5 (Experimental): Buprenorphine + Rifampin
  Interventions: Drug: Rifampin; Drug: Buprenorphine
- 6 (Experimental): Buprenorphine + Rifabutin
  Interventions: Drug: Rifabutin; Drug: Buprenorphine

INTERVENTIONS:
Drug: Fosamprenavir/Ritonavir — 1400/200 mg once daily for 15 days total
  Other Names: Lexiva/Norvir
  Arms: 1; 2
Drug: Darunavir/Ritonavir — 800/100 mg once daily for 15 days total
  Other Names: Prezista/Norvir
  Arms: 3; 4
Drug: Rifampin — 600 mg once daily for 15 days total
  Arms: 5
Drug: Rifabutin — 300 mg once daily for 15 days total
  Arms: 6
Drug: Buprenorphine — FOSAMPRENAVIR/RITONAVIR Dosing information: 1400 mg fosamprenavir + 200 mg ritonavir once daily for 15 days
  DARUNAVIR/RITONAVIR Dosing information: 800 mg darunavir + 100 mg ritonavir once daily for 15 days
  RIFAMPIN Dosing information: 600 mg once daily in the morning for 15 days
  RIFABUTIN Dosing information: 300 mg once daily in the morning for 15 days
  Other Names: Suboxone
  Arms: 1; 3; 5; 6

SUMMARY:
The purpose of this study is to examine the interactions of buprenorphine-naloxone, a medication used to treat opiate (heroin or prescription narcotic) dependence, and medications used in the treatment of HIV disease including atazanavir (Reyataz), fosamprenavir (Lexiva), didanosine (Videx), tenofovir (Viread), atazanavir (Reyataz)/ritonavir (Norvir), fosamprenavir (Lexiva)/ritonavir (Norvir), lamivudine (Epivir), or darunavir (please note that we have completed drug interaction studies for buprenorphine with atazanavir, atazanavir/ritonavir, didanosine, tenofovir and lamivudine) at the PI's previous university; for this CHR application only the studies needed to be completed at UCSF/SFGH will be discussed) or tuberculosis(TB) (rifampin or rifabutin) medications (note: supplement application currently pending). Participants are those with opioid dependence who qualify for buprenorphine/naloxone treatment or they are healthy subjects without opioid dependence who participate in pharmacokinetics studies of the antiretroviral medications. A total of 160 such individuals will be enrolled in these studies (please note that the studies have been ongoing at Virginia Commonwealth University for 3 years so that the total number of participants to be recruited at UCSF/SFGH will be about 50 protocol completers). Participants take the HIV or tuberculosis medicine(s) for up to 15 days (depending on the medication(s) administered and ability to schedule blood and urine sampling sessions).

DETAILED DESCRIPTION:
The overall objective of this project, RO1 DA 13004 "Opioids and HIV Medications: Interactions in Drug Abusers" and the supplement "Interaction of Buprenorphine and TB Medications," is to continue to improve the clinical care of human immunodeficiency virus (HIV)-infected, substance-abusing patients by identifying significant interactions that may occur between drugs commonly used to treat HIV disease or tuberculosis and buprenorphine, the newest opioid used for maintenance treatment of opioid dependence and an important addition to existing substance abuse pharmacotherapies because its use is not restricted to specialized opiate treatment programs. The research funded by this grant over the past years has shown the presence of significant and clinically important drug interactions between methadone and LAAM in combination with antiretroviral medications. Understanding these drug interactions will allow physicians to safely and more effectively treat HIV disease in opioid-dependent patients. The following specific aims are yet to be completed for this project which has another 2 years of a 5 year funding period: 1. Continuation of studies to determine whether the pharmacokinetics of buprenorphine are affected by coadministration of any of the following HIV medications fosamprenavir/ritonavir, darunavir or the TB medications, rifampin or rifabutin. This will be done by comparing the pharmacokinetics of buprenorphine in the absence and presence of each HIV medication using a within subjects study design with participants who are opioid-dependent, without HIV infection, and receiving medication maintenance treatment with buprenorphine/naloxone (please note that naloxone absorption is negligible and is added to the buprenorphine preparation by the drug manufacturer to diminish the likelihood of diversion of the drug to injected abuse). These studies will allow an answer to a major question of concern to patients and their clinicians: Could starting one of these HIV medications or TB medications result in opioid overdose or withdrawal? These studies will determine whether buprenorphine accumulation and toxicity might occur or whether buprenorphine concentrations at standard medication doses will be subtherapeutic and/or expose the patient to the risk of opioid withdrawal symptoms during conjoint HIV or TB therapy. 2. Continuation of studies to determine whether the pharmacokinetics of the HIV medications fosamprenavir/ritonavir or darunavir, are affected by coadministration of buprenorphine. This will be done in between-subjects studies by comparing the pharmacokinetics of each HIV medication in groups of patients treated with buprenorphine and in a control group without opioid dependence or HIV infection. It will be important to identify any interaction leading to increased exposure to an HIV therapeutic with a concomitant increase in side-effects and toxicities. In addition to unnecessary discomfort and hazard, this may lead to non-adherence and/or increased substance abuse particularly if side effects are interpreted as opioid withdrawal. Equally important, substantial decreases in levels of HIV drugs could lead to subtherapeutic levels, inadequate viral suppression, and the development of antiretroviral resistance and therapeutic failure. (Please note that for the TB medications supplemental studies only the within-subjects component with buprenorphine will be completed due to budgetary constraints of the supplement.) Important clinical effects related to concomitant buprenorphine/HIV therapeutic or TB medication administration are also collected including: 1. Measures of opioid withdrawal symptoms will be collected prior to and following simultaneous buprenorphine/antiretroviral administration 2. Measures of cognitive function will be collected prior to and following simultaneous buprenorphine/antiretroviral administration 3. Measures of the occurrence of adverse events will be systematically collected and chronicled prior to and following simultaneous buprenorphine/antiretroviral administration 4. Effect of buprenorphine alone and buprenorphine in combination with antiretroviral administration on cardiac conduction will be obtained with serial electrocardiograms. 5. Effect of buprenorphine alone and in combination with antiretroviral or anti-TB medication administration on hepatic function through serial collection of laboratory blood tests of liver function to gain insight into the potential of these drugs to produce hepatotoxicity. The experimental protocol allows both sets of studies (Aims 1 and 2) to be accomplished simultaneously in the same buprenorphine-maintained subjects, thereby achieving substantial efficiencies in the current project. The studies offer a cost-effective method for rapid determination of the presence and clinical significance of drug interactions between buprenorphine and pharmacotherapies for infectious diseases of great clinical importance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be in good health as determined by a physical examination and screening laboratory tests and urinalysis, and will meet the criteria of opioid dependence, but will not be physiologically dependent on any other drugs or alcohol; those with history of current binge alcohol use will also be excluded. Subjects will be enrolled in buprenorphine treatment and must be on a stable, standard clinical dose (4-20 mg/d) for at least 2 weeks prior to initiation of pharmacokinetics study.
* Control subjects who are non-opioid dependent, are not physiologically dependent on any other drugs or alcohol and volunteer for the HIV medications pharmacokinetics studies alone must be in good health as determined by a physical examination and screening laboratory studies as described below.
* Age 18 or older.
* Able to give voluntary, signed, informed consent.

Exclusion Criteria:

* Patients who are receiving concurrently other drugs that are inducers or inhibitors of hepatic microsomal enzymes.
* Patients with a known sensitivity to the HIV therapeutics to be studied.
* Pregnant women or nursing mothers. All women who are sexually active and capable of becoming pregnant must have a negative pregnancy test within one week prior to entry into these studies.
* Major psychotic illness or suicidality.
* Clinically active hepatitis (primarily Hepatitis B or C in opioid dependent subjects) with liver enzyme elevations > 3 times the upper limit of normal
* Those with diabetes, hyperlipidemia, coagulation disorders, or renal disease will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Effect of ARV or Tuberculosis Medication on Buprenorphine | 2007-2010

CONTACTS AND LOCATIONS:
Overall Officials: Elinore F McCance-Katz, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States